CLINICAL TRIAL: NCT06599242
Title: The Effects of Basic Body Awareness Therapy on Balance, Jumping Performance and Sports Injury Anxiety in American Football Players
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: YeditepeU-PTR-AEA-01
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-06

CONDITIONS: Sport Injury
Keywords: American Football; Basic Body Awareness Therapy,

STUDY DESIGN:
Intervention Model Description: Athletes who play American football at Yeditepe University American Football Team Club and volunteered to participate in the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Basic Body Awareness Therapy Group ( BBATG) (Experimental): Basic Body Awareness Therapy Exercises American football team training
  Interventions: Other: Basic Body Awareness Therapy; Other: American football team training
- Control Group (Active Comparator): American football team training
  Interventions: Other: American football team training

INTERVENTIONS:
Other: Basic Body Awareness Therapy — Basic Body Awareness Therapy is an exercise approach belonging to physiotherapists
  Arms: Basic Body Awareness Therapy Group ( BBATG)
Other: American football team training — American football team training

SUMMARY:
This study aims to investigate the effects of Basic Body Awareness Therapy (BBAT) on balance, jump performance and sports injury anxiety in American football players. Participants were divided into two groups, Body Awareness Therapy Treatment Group (n=22) and a Control group(n=22), by computer-based randomization.

DETAILED DESCRIPTION:
This study aims to investigate the effects of Basic Body Awareness Therapy (BBAT) on balance, jump performance and sports injury anxiety in American football players. Participants were divided into two groups, Body Awareness Therapy Treatment Group (n=22) and a Control group(n=22), by computer-based randomization. Before starting the study, all participants were given detailed information about the content of the study and filled out a voluntary consent form. All participants in both groups were evaluated under the same conditions and surveys were conducted. The intervention group was given BBAT exercises by a physiotherapist who had received BBTA training 2 days a week for 6 weeks. All participants continued their team training during this period. At the end of the 6 weeks, all participants were given the same conditions and the surveys were repeated.

ELIGIBILITY:
Inclusion Criteria:

* Being a licensed American football player
* Playing in the university league
* Continue training for at least 1 year
* To be between the ages of 18-25
* Volunteering to participate in the study
* No disabilities for assessment tests

Exclusion Criteria:

* Orthopedic injury in the last 6 months
* Having undergone lower extremity surgery in the last 1 year
* Loss of vision and hearing
* Presence of a neurological defect- The athlete (if female) is not pregnant

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2024-06-03 (Actual); Primary Completion 2024-09-16 (Estimated); Study Completion 2024-09-16 (Estimated)

PRIMARY OUTCOMES:
Balance | 6 weeks
  Static balance ( Flamingo Balance Test) and dynamic balance ( Y Balance Test )

SECONDARY OUTCOMES:
Jump Performance | 6 weeks
  Vertical and Horizontal Jump Test are used

OTHER OUTCOMES:
Sports Injury Anxiety | 6 weeks
  Sports Injury Anxiety Scale is used
Body Awareness Questionnaire | 6 weeks
  Body Awareness Questionnaire is used

CONTACTS AND LOCATIONS:
Locations (1):
- Yeditepe University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No